CLINICAL TRIAL: NCT02843204
Title: Combination of Anti-PD-1 and NK Immunotherapy for Recurrent Solid Tumors
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Fuda Cancer Hospital, Guangzhou (Other)
Collaborators: Shenzhen Hank Bioengineering Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NK-PD-1
Record Dates: First submitted 2016-07-21; First posted 2016-07-25 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Malignant Solid Tumour
Keywords: Solid tumor; Anti-PD-1; NK immunotherapy
MeSH Terms: interventions — pembrolizumab

ARMS (2):
- Pembrolizumab and NK immunotherapy (Experimental): In this group, the patients will receive regular Pembrolizumab first to control tumor burden; then NK immunotherapy will be given. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Drug: Pembrolizumab; Biological: NK immunotherapy
- Pembrolizumab (Active Comparator): In this group, the patients will receive regular Pembrolizumab to control tumor burden. The check indexes are CT scan and blood tests (including tumor markers, lymphocyte subsets and circulating tumor cell).
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Patients received i.v. pembrolizumab (10 mg/kg) on day 1 of a 21-day cycle, until disease progression, discontinuation due to unacceptable toxicity, withdrawal of consent or study closure
  Other Names: Keytruda
Biological: NK immunotherapy — Each treatment: about 10 billion cells in all, infusion in 3 times, i.v.
  Arms: Pembrolizumab and NK immunotherapy

SUMMARY:
The aim of this study is the safety and efficacy of anti-PD-1 plus NK immunotherapy to multiple solid tumors.

DETAILED DESCRIPTION:
By enrolling patients with solid tumors adapted to enrolled criteria, this study will document for the first time the safety and the short and long term efficacy of the combined therapy using anti-PD-1 and natural killer (NK) cells.

The safety will be evaluated by statistics of adverse reactions. The efficacy will be evaluated according to local relief degree, progress free survival (PFS) and overall survival (OS).

ELIGIBILITY:
Inclusion Criteria:

* All standard therapies have failed according to NCCN guidelines or the patient refuses standard therapies after cancer recurrence
* Progression after chemotherapy or appropriate TKI treatment for those patients with an EGFR-sensitizing mutation or ALK rearrangement
* KPS ≥ 70, lifespan > 3 months, PD-L1 TPS of 1% or greater
* Platelet count ≥ 80×10^9/L，white blood cell count ≥ 3×10^9/L, neutrophil count ≥ 2×10^9/L, hemoglobin ≥ 80 g/L

Exclusion Criteria:

* Patients with cardiac pacemaker
* Patients with brain metastasis
* Patients with grade 3 hypertension or diabetic complication, severe cardiac and pulmonary dysfunction, myelosuppression, autoimmune disease, pneumonitis
* Previous treatment with a therapeutic antibody against CTLA4, PD-L1, or PD-1, or PD-L1/PD-1 pathway-targeting agents.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2017-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
PFS | 2 year
  PFS was defined as the interval between treatment initiation and local relapse,
OS | 3 years
  OS was calculated as the interval from treatment initiation to death.

SECONDARY OUTCOMES:
PD-1 | 3 months
  Peripheral blood (6 mL) was obtained from healthy donors and patients before treatment and 90 days after treatment for the detection of PD-1
Tumor size | 3 months
  The tumor responses of the enrolled patients were assessed by CT in accordance with RECIST v1.1.Institute Common Terminology Criteria for Adverse Events (v4.0).
CEA | 3 months
  CEA was evaluated by a chemiluminescent immunoassay before treatment and 90 days after treatment.
CTC | 3 months
  The absolute number of CD45-CK+ CD326+ cells was used to quantitate the CTC levels.

CONTACTS AND LOCATIONS:
Overall Officials: Jibing Chen, MD, PhD, Principal Investigator — Fuda Cancer Hospital, Guangzhou
Locations (1):
- Cancer Institute in Fuda Cancer Hospital, Guangzhou, Guangdong, China

REFERENCES:
- [Derived] Lin M, Luo H, Liang S, Chen J, Liu A, Niu L, Jiang Y. Pembrolizumab plus allogeneic NK cells in advanced non-small cell lung cancer patients. J Clin Invest. 2020 May 1;130(5):2560-2569. doi: 10.1172/JCI132712. PMID 32027620